CLINICAL TRIAL: NCT02828735
Title: REspiration Patterns in REVEAL LINQ Insertable Cardiac Monitor
Brief Title: Respiration Patterns With Impedance in LINQ
Acronym: EPIQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic BRC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EPIQ
Record Dates: First submitted 2015-07-20; First posted 2016-07-12 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Respiration assessment (Other)
  Interventions: Device: respiration assessment

INTERVENTIONS:
Device: respiration assessment — Respiration Breathing Exercise

SUMMARY:
The purpose of the study is to evaluate the use of subcutaneous impedance measured with an implanted Medtronic Reveal LINQ™ insertable cardiac monitor (ICM) as respiratory rate monitor.

ELIGIBILITY:
Inclusion Criteria:

* Suspected arrhythmia Diastolic Heart Failure and/or in Renal Failure.
* Chronic Kidney Disease (CKD) in Stage 5 (GFR = <15 mL/min).
* Diastolic Heart Failure in class II and class III (class IV to be considered in end stage and non-reversible).
* Willing to sign the informed consent form.
* Greater than 18 years of age.

Exclusion Criteria:

* Enrolled in another study that could confound the results of this study, without documented pre-approval from a Medtronic study manager.
* Significant respiratory diseases such as COPD or pulmonary hypertension.
* Frequent arrhythmias, including PVC's.
* Known systolic heart failure.
* Recent infection.
* Allergenic or rejection reaction to materials used in incision/insertion tools, Reveal LINQ™ ICM exterior or incision closure method.
* Active implanted cardiac medical device (e.g. IPG, ICD, CRT, etc).
* Not suitable for Reveal LINQ™ implantation (e.g., severe cachexia, dermatologic conditions of the skin) or any concomitant condition which in the opinion of the investigator would not allow a safe participation in the study.
* Body conditions that would complicate accurate measurement of respiratory efforts with an external device deployed around the chest.
* Not able to take the postures as necessary for the study protocol and not able to walk continuously for a period of 6 minutes.
* Any concomitant condition which in the opinion of the investigator would not allow a safe participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
feasibility of respiration detection | up to 18 months
  Respiratory Maneuvers and Device interrogation

CONTACTS AND LOCATIONS:
Overall Officials: Mpiko Ntsekhe, Principal Investigator — Groote Schuur Hospital, Cape Town, South Africa
Locations (1):
- Groote Schuur Hospital, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Undecided